CLINICAL TRIAL: NCT03464448
Title: Mechanistic Studies of Teriflunomide in Relapsing Remitting Multiple Sclerosis: Regulatory B Lymphocytes as Central Mediators of the Therapeutic Effects of Teriflunomide in MS
Brief Title: Mechanistic Studies of Teriflunomide in RRMS
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yang Mao-Draayer, Professor of Neurology, University of Michigan
Other Study IDs: HUM00136966
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Teriflunomide; B cell; T cell; cytokines
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — teriflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected after 3, 6, 9, 12, 18 and 24 months of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Patients with RRMS who have been newly prescribed Teriflunomide.
  Interventions: Drug: Teriflunomide
- 2: Healthy Controls

INTERVENTIONS:
Drug: Teriflunomide — AUBAGIO® (teriflunomide) is a prescription medicine used to treat relapsing forms of multiple sclerosis (MS), which inhibits pyrimidine de novo synthesis by blocking the enzyme dihydroorotate dehydrogenase.
  Other Names: Aubagio
  Groups: 1

SUMMARY:
This study is to address the mechanism of action of teriflunomide in a phase IV open label trial with Teriflunomide in multiple sclerosis. Researchers will recruit 20 relapsing remitting multiple sclerosis patients (Group 1) start on treatment with teriflunomide (Aubagio). Patients will be enrolled from the Multiple Sclerosis Center at the University of Michigan Health System in Ann Arbor. Meanwhile, 10 healthy controls will be recruited, to establish a healthy baseline for B and T cells, which are affected by both MS and its treatment (Group 2). This Study will collect baseline pre-treatment blood samples periodically for up to 2 years. Blood biomarker changes will be correlated with clinical response to teriflunomide treatment intervention.

DETAILED DESCRIPTION:
Multiple sclerosis is the most common autoimmune inflammatory and debilitating chronic demyelinating disease of the central nervous system mainly affecting young adults. There is a tremendous need to understand the mechanism of action of the treatment and how they might work in multiple sclerosis patients. Most recently, teriflunomide (AubagioTM) has been demonstrated to act as an immune modulatory therapy for patients with multiple sclerosis. Although one biochemical mechanism of action is understood to be related to inhibition of dihydroorotate dehydrogenase (DHODH) which affects synthesis of pyrimidine nucleotides, there have also been reports that the functions of regulatory T cells are promoted by these drugs independent of DHODH. Much accumulating evidence suggests that specialized subsets of B lymphocytes are important inducers of regulatory T cells, as well as having killer functions that may preferentially target TH1 and TH17 cells.

This study aims to address the mechanism of action of teriflunomide in a phase IV open label trial with Teriflunomide in multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically-defined relapsing-remitting MS (RRMS) who " are newly starting on teriflunomide (AubagioTM) at the time of enrollment " have no evidence of relapse or corticosteroid treatment use within 2 months prior to enrollment

   OR

   Healthy controls who do not have a significant medical condition such as cancer, chronic infection, or autoimmune disease, have not taken steroids in the past 2 months, and who are not on an immune suppressant medication.
2. Ability to give informed consent
3. Willing to have blood drawn as scheduled in the protocol
4. Willing and able to complete all procedures and evaluations related to the study

Exclusion Criteria:

1. Medical or psychiatric conditions that may affect the patient's ability to give informed consent
2. Has received an experimental drug within 30 days of enrollment
3. Concomitant other disease modifying medications (such as Rebif, Betaseron, Avonex, Copaxone, Gilenya, Tecfidera, Alemtuzumab, methotrexate, azathioprine, mitoxantrone, cyclophosphamide, cyclosporine, natalizumab, rituxan, ocrelizumab, etc.) without the minimal washout period stated below:

   " rebif, betaseron, avonex, copaxone within 1 month " zinbryta, plegridy, gilenya, tecfidera within 2 months " natalizumab within 3 months " immunosuppressive/chemotherapeutic medications (e.g. azathioprine, methotrexate) within 6 months " cyclophosphamide within 1 year " rituximab, ofatumumab, ocrelizumab, cladribine within 1 year " alemtuzumab at any time " any mitoxantrone during previous 2 years prior to randomization or evidence of cardiotoxicity following mitoxantrone or a cumulative life-time dose of more than 60 mg/m2 " lymphoid irradiation, bone marrow transplantation or other immunosuppressive treatments with effects potentially lasting over 6 months, at any time
4. Has any contraindication to high-dose immunotherapy, including pregnancy, trying to become pregnant, or breast feeding during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 20 multiple sclerosis (MS) patients and 10 healthy controls will be recruited to voluntarily donate blood for the study. Blood samples will be collected prior to starting teriflunomide treatment (baseline) and after 3, 6, 9, 12, 18 and 24 months of treatment (+/- 2 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of regulatory and effector B cell subset | From baseline to 6 months and 12 months
  Compare aubagio treatment to baseline and to healthy controls

SECONDARY OUTCOMES:
Change in frequency of CD4+ Th17, Th1, Th2, and Treg cells | From baseline to 6 months and 12 months
  Compare aubagio treatment to baseline and to healthy controls
Change in chemokine levels | From baseline to 6 months and 12 months
  Compare aubagio treatment to baseline and to healthy controls
Change in cytokine levels | From baseline to 6 months and 12 months
  Compare aubagio treatment to baseline and to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mao-Draayer, MD/PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser SL, Oksenberg JR. The neurobiology of multiple sclerosis: genes, inflammation, and neurodegeneration. Neuron. 2006 Oct 5;52(1):61-76. doi: 10.1016/j.neuron.2006.09.011. PMID 17015227
- [Background] Trapp BD, Nave KA. Multiple sclerosis: an immune or neurodegenerative disorder? Annu Rev Neurosci. 2008;31:247-69. doi: 10.1146/annurev.neuro.30.051606.094313. PMID 18558855
- [Background] Bar-Or A, Pachner A, Menguy-Vacheron F, Kaplan J, Wiendl H. Teriflunomide and its mechanism of action in multiple sclerosis. Drugs. 2014 Apr;74(6):659-74. doi: 10.1007/s40265-014-0212-x. PMID 24740824
- [Background] Lundy SK, Wu Q, Wang Q, Dowling CA, Taitano SH, Mao G, Mao-Draayer Y. Dimethyl fumarate treatment of relapsing-remitting multiple sclerosis influences B-cell subsets. Neurol Neuroimmunol Neuroinflamm. 2016 Mar 3;3(2):e211. doi: 10.1212/NXI.0000000000000211. eCollection 2016 Apr. PMID 27006972
- [Background] Claussen MC, Korn T. Immune mechanisms of new therapeutic strategies in MS: teriflunomide. Clin Immunol. 2012 Jan;142(1):49-56. doi: 10.1016/j.clim.2011.02.011. Epub 2011 Mar 1. PMID 21367665
- [Background] Baban B, Liu JY, Mozaffari MS. Aryl hydrocarbon receptor agonist, leflunomide, protects the ischemic-reperfused kidney: role of Tregs and stem cells. Am J Physiol Regul Integr Comp Physiol. 2012 Dec;303(11):R1136-46. doi: 10.1152/ajpregu.00315.2012. Epub 2012 Oct 24. PMID 23100028
- [Background] Korn T, Magnus T, Toyka K, Jung S. Modulation of effector cell functions in experimental autoimmune encephalomyelitis by leflunomide--mechanisms independent of pyrimidine depletion. J Leukoc Biol. 2004 Nov;76(5):950-60. doi: 10.1189/jlb.0504308. Epub 2004 Aug 24. PMID 15328336
- [Background] Weigmann B, Jarman ER, Sudowe S, Bros M, Knop J, Reske-Kunz AB. Induction of regulatory T cells by leflunomide in a murine model of contact allergen sensitivity. J Invest Dermatol. 2006 Jul;126(7):1524-33. doi: 10.1038/sj.jid.5700228. Epub 2006 Mar 16. PMID 16543898
- [Background] Carter NA, Rosser EC, Mauri C. Interleukin-10 produced by B cells is crucial for the suppression of Th17/Th1 responses, induction of T regulatory type 1 cells and reduction of collagen-induced arthritis. Arthritis Res Ther. 2012 Feb 8;14(1):R32. doi: 10.1186/ar3736. PMID 22315945
- [Background] Flores-Borja F, Bosma A, Ng D, Reddy V, Ehrenstein MR, Isenberg DA, Mauri C. CD19+CD24hiCD38hi B cells maintain regulatory T cells while limiting TH1 and TH17 differentiation. Sci Transl Med. 2013 Feb 20;5(173):173ra23. doi: 10.1126/scitranslmed.3005407. PMID 23427243
- [Background] Iwata Y, Matsushita T, Horikawa M, Dilillo DJ, Yanaba K, Venturi GM, Szabolcs PM, Bernstein SH, Magro CM, Williams AD, Hall RP, St Clair EW, Tedder TF. Characterization of a rare IL-10-competent B-cell subset in humans that parallels mouse regulatory B10 cells. Blood. 2011 Jan 13;117(2):530-41. doi: 10.1182/blood-2010-07-294249. Epub 2010 Oct 20. PMID 20962324
- [Background] Mann MK, Maresz K, Shriver LP, Tan Y, Dittel BN. B cell regulation of CD4+CD25+ T regulatory cells and IL-10 via B7 is essential for recovery from experimental autoimmune encephalomyelitis. J Immunol. 2007 Mar 15;178(6):3447-56. doi: 10.4049/jimmunol.178.6.3447. PMID 17339439
- [Background] Matsushita T, Horikawa M, Iwata Y, Tedder TF. Regulatory B cells (B10 cells) and regulatory T cells have independent roles in controlling experimental autoimmune encephalomyelitis initiation and late-phase immunopathogenesis. J Immunol. 2010 Aug 15;185(4):2240-52. doi: 10.4049/jimmunol.1001307. Epub 2010 Jul 12. PMID 20624940
- [Background] Ray A, Basu S, Williams CB, Salzman NH, Dittel BN. A novel IL-10-independent regulatory role for B cells in suppressing autoimmunity by maintenance of regulatory T cells via GITR ligand. J Immunol. 2012 Apr 1;188(7):3188-98. doi: 10.4049/jimmunol.1103354. Epub 2012 Feb 24. PMID 22368274
- [Background] Klinker MW, Lundy SK. Multiple mechanisms of immune suppression by B lymphocytes. Mol Med. 2012 Feb 10;18(1):123-37. doi: 10.2119/molmed.2011.00333. PMID 22033729
- [Background] Cross AH, Stark JL, Lauber J, Ramsbottom MJ, Lyons JA. Rituximab reduces B cells and T cells in cerebrospinal fluid of multiple sclerosis patients. J Neuroimmunol. 2006 Nov;180(1-2):63-70. doi: 10.1016/j.jneuroim.2006.06.029. Epub 2006 Aug 14. PMID 16904756